CLINICAL TRIAL: NCT07355413
Title: Frailty, Geriatric Syndromes and Care Pathways of Older Adults Living With HIV in West Africa
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 0496s FraGericare-WA
Record Dates: First submitted 2026-01-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Older Adults
Keywords: HIV; Frailty; Geriatric syndromes; Care pathways
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV positive group: Individuals aged 60 years and over living with HIV-1 and/or HIV-2 attending HIV care centers in Abidjan, Bobo-Dioulasso and Lomé.
- HIV negative group: Individuals aged 60 years and over without HIV, matched by sex and age group.

SUMMARY:
With currently available antiretroviral therapy, people living with HIV (PLWHIV) are living longer. This exposure to HIV and combination antiretroviral therapy may accelerate the aging of this population, thus increasing the prevalence of premature frailty.

There are few data on the prevalence of frailty and geriatric syndromes among older people living with HIV (OpHIV) in sub-Saharan Africa (SSA) and the screening and diagnostic tools to identify them.

The initiation contract financed by the ANRS-MIE in 2021 whose objective was to 1) carry out an inventory and evaluate the feasibility of a project for monitoring OpHIV in Burkina-Faso in Côte d'Ivoire and Togo and 2) to select the collection tools adapted to the description of geriatric syndromes in these elderly people has allowed to highlight the following (i) The collection of data on geriatric conditions and syndromes is almost non-existent in the daily care and management practice (ii) there is a significant proportion (10,6%) of PLWHIV aged 60 years and over in the active files of the PLWHIV care centers that participated in the survey (iii) Adapted screening tools have been selected and will allow documentation of the above-mentioned syndromes. This research project, which follows on from this initiation contract, will therefore make it possible to obtain data from the geriatric evaluation, to identify the specificities of PLWHIV by comparing them to a population not infected with HIV and to propose geriatric management adapted to PLWHIV. Its innovative nature also lies in its mixed approach combining quantitative and qualitative methods, which will make it possible to document the needs and resources for the care of PLWHIV in a global and holistic manner.

600 participants, aged 60 years and over (300 living with HIV and 300 not living with HIV), in three West African countries (Burkina Faso, Côte d'Ivoire, Togo) will be included in this study whose primary objective is to compare the prevalence of frailty among people aged 60 years and over (PA60) between HIV-infected and non-HIV-infected; the secondary objective is to estimate the prevalence of frailty among PA60 according to HIV status. A population-based matching will be performed on sex and age class (threshold 70 years), during the recruitment of HIV- PA60.

This will be a mixed study combining:

* A "clinical" component comprising a stratified, comparative, international, multicenter cross-sectional study;
* A "health systems strengthening" component combining a quantitative cross-sectional survey and a qualitative survey;
* A qualitative socio-anthropological component including individual interviews and focus groups with people living with HIV60, their families and caregivers.

The 3 components will be conducted with a time lag between the different components due to the overlapping constitution of the source populations.

Most research on aging with HIV in the context of SSA has been very clinically focused (e.g., frailty or cognitive impairment). This research will provide a more comprehensive approach that takes into account the different levels of factors influencing health (individual, health system, social environment).

DETAILED DESCRIPTION:
Methodology:

This is a mixed study combining:

* a "clinical" component comprising a comparative, international, multicenter, two-strata (HIV+ and HIV-) cross-sectional study;
* a "social sciences" component combining a quantitative cross-sectional survey and a qualitative survey involving individual interviews and focus groups with PA60, their families and caregivers.

Interventions:

* Screening for several comorbidities (high blood pressure, diabetes, dyslipidemia, kidney failure, undernutrition, depression).
* Comprehensive management including prevention strategies adapted to the various comorbidities mentioned above and their complications.

Statistical method:

Use of mixed approaches. For quantitative indicators, descriptive analysis techniques, bivariate analysis (Student t test or Wilcoxon test for quantitative variables, Chi² or Fisher test for categorical variables) and multivariate analysis (logistic regression).

ELIGIBILITY:
Inclusion Criteria:

* HIV+ Group

  * Person 60 years of age and older
  * Infected with HIV-1 and/or 2
  * Able to move around the data collection site
  * Having given free and informed consent
* HIV- Group

  * Person 60 years of age and older
  * HIV-uninfected
  * Able to move around the data collection site
  * Having given free and informed consent

Exclusion Criteria:

Person deprived of liberty (guardianship, curatorship, judicial safeguard) Karnofsky Index 50≤50% Hospitalized

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical component
  The targets of this component of the study are two specific populations:
  * People over the age of 60 (PA60) infected with HIV who are receiving treatment at HIV care centers in Abidjan (Ivory Coast), Bobo-Dioulasso (Burkina Faso), and Lomé (Togo), or who have recently been infected with HIV;
  * People over the age of 60 who are not infected with HIV.
  Social science component:
  * PA60 HIV+/HIV-
  * Caregivers
  * Healthcare providers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of frailty by HIV status among people aged 60 years and older (PA60) in West Africa | At 12 months

SECONDARY OUTCOMES:
Prevalence of frailty in AP60 | At 12 months
Number and proportion of AP60 with geriatric syndrome | At 12 months
  Including cognitive, visual and hearing disorders, depression, undernutrition, dehydration, pain, urinary and fecal continence disorders, gait and balance disorders, according to HIV status
Number and proportion of AP60 with at least one comorbidity | At 12 months
  Including cancer, dyslipidemia, diabetes, hypertension, history of myocardial infarction or stroke, osteoarticular disease, renal failure, according to HIV status
Factors associated with the presence of geriatric syndromes | At t12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde ALLAVENA, Principal Investigator — Nantes University Hospital; Raoul MOH, Principal Investigator — Programme PAC-CI CHU de Treichville
Locations (6):
- Hôpital de jour du CHU Sourou Sanou, Bobo-Dioulasso, Burkina Faso
- Côte d’Ivoire (3):
  - Centre Médical de Suivi des donneurs de sang (CMSDS), Treichville, Abidjan Autonomous District
  - Service des Maladies Infectieuses et Tropicales (SMIT), Treichville, Abidjan Autonomous District
  - Centre de Prise en Charge de Formation et de Recherche (CEPREF), Yopougon, Abidjan Autonomous District
- Togo (2):
  - ONG Espoir Vie Togo, Lomé
  - Service des Maladies Infectieuses et Tropicales-CHU Sylvanus Olympio, Lomé